CLINICAL TRIAL: NCT00569309
Title: Immune Reconstitution After Autologous Hematopoietic Stem Cell Transplantation for High-Risk Lymphoma and Myeloma
Brief Title: Immune Reconstitution After Autologous Hematopoietic Stem Cell Transpl for High-Risk Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07044
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Small Intestine Cancer
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent adult Hodgkin lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; adult nasal type extranodal NK/T-cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; small intestine lymphoma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Hodgkin Disease; Lymphoma, Extranodal NK-T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevnar (Experimental): The conjugate vaccine for Streptococcus pneumoniae will be administered during weeks 9, 17, and 25 after autologous HSCT - the study nurse will arrange for the vaccine to be administered at the specified time and the patient will be instructed to notify an investigator or study nurse of any side effects of vaccine administration. At the specified times, patients will fill out the quality-of-life assessment. All patients enrolled on this trial will have samples procured for all proposed laboratory correlative studies.
  Interventions: Biological: Streptococcus pneumoniae; Other: laboratory correlative studies; Other: quality-of-life assessment

INTERVENTIONS:
Biological: Streptococcus pneumoniae — Patients will receive 0.5 mL Prevnar in the deltoid muscle during weeks 9, 17, and 25 after autologous hematopoietic stem cell transplantation (HSCT)
  Other Names: Prevnar; PCV7
Other: laboratory correlative studies — Approximately 30-mL of blood will be collected and sent to the appropriate research lab(s) for processing.
  Other Names: laboratory biomarker analysis; blood samples
Other: quality-of-life assessment — Responses to Hospital Anxiety and Depression Scale, 9-item brief fatigue inventory 57, brief pain inventory, and the FACT-G. This should take each patient approximately 10-15 minutes to fill out all these surveys per instance.
  Other Names: QOL

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill cancer cells. Giving vaccine therapy after an autologous stem cell transplant may kill any cancer cells that remain after transplant.

PURPOSE: This clinical trial is studying how well vaccine therapy works in treating patients who have undergone autologous stem cell transplant for high-risk lymphoma or multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess immune reconstitution as measured by response to pneumococcal polyvalent vaccine, NK-cell activity against autologous lymphoblastoid cell lines, and cytomegalovirus and Epstein-Barr virus tetramer responses in patients who have undergone autologous hematopoietic stem cell transplantation for high-risk lymphoma or multiple myeloma.

Secondary

* Assess the absolute number of circulating regulatory T-cells and the function of these cells as measured by their expression of TGFβ and interleukin-10 (IL-10).
* Evaluate the effect of conditioning therapy on quality of life, including functional status, fatigue, and depression, in these patients.
* Correlate quality of life with inflammatory cytokine production of peripheral blood monocytes at specified time points.
* Provide baseline immune reconstitution and quality of life pilot data for comparison in future post-transplant immunotherapy trials.

OUTLINE: Patients receive pneumococcal polyvalent vaccine intramuscularly once in weeks 9, 17, and 25 after autologous hematopoietic stem cell transplantation.

Blood samples are collected periodically for correlative and immunological studies.

Quality of life (QOL) is assessed periodically using the QOL short form (SF-36, 4-week version), the Center for Epidemiologic Studies Depression scale (CES-D), and the Multidimensional Fatigue Symptom Inventory (MFSI-30).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma OR any of the following high-risk lymphomas:

  * Diffuse large B-cell lymphoma meeting any of the following criteria:

    * Failed induction therapy but responded to salvage therapy
    * Relapsed < 1 year after completion of induction therapy
    * Elevated lactic dehydrogenase (LDH) at relapse
    * Stage III or IV disease at relapse
    * Positive PET scan after induction or salvage therapy
    * Age 60 to 75 years
  * Follicular lymphoma meeting any of the following criteria:

    * Progressive disease after two or more prior regimens
    * Transformed to aggressive diffuse large B-cell lymphoma but is still chemotherapy sensitive
    * Not considered to be a good candidate for allogeneic stem cell transplantation
  * Hodgkin lymphoma meeting any of the following criteria:

    * Primary refractory disease
    * Relapsed < 1 year after completion of induction therapy
    * Relapsed with PET positive disease after salvage therapy
    * Relapsed refractory disease and is not considered to be a good candidate for allogeneic stem cell transplantation
  * Mantle cell lymphoma meeting any of the following criteria:

    * Chemotherapy sensitive disease after induction therapy
    * Chemotherapy sensitive relapsed disease and is not considered to be a good candidate for allogeneic stem cell transplantation
  * T-cell non-Hodgkin lymphoma (NHL) meeting any of the following criteria:

    * Peripheral T-cell lymphoma, not otherwise specified meeting at least one of the following criteria:

      * High LDH at diagnosis
      * Marrow involvement at diagnosis
      * Age > 60 years at diagnosis
      * Low platelet count at diagnosis
      * Chemotherapy sensitive relapsed disease
    * Angioimmunoblastic lymphadenopathy with dysproteinemia
    * ALK-negative anaplastic NHL
    * Enteropathy-associated T-cell NHL
    * Stage III or IV NK-/T-cell NHL at diagnosis
    * NK-blastic NHL
* Has undergone autologous hematopoietic stem cell transplantation and received 200 mg/m² of melphalan (for multiple myeloma) OR BEAM chemotherapy comprising carmustine, etoposide, cytarabine, and methotrexate (for high-risk lymphoma) as conditioning therapy

PATIENT CHARACTERISTICS:

* ECOG or WHO performance status 0-2
* ANC ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 1.5 mg/dL
* Alkaline phosphatase ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 2 times the ULN
* Not pregnant or nursing
* No severe or uncontrolled systemic illness
* No "currently active" second malignancy, other than nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Patients are not considered to have a "currently active" malignancy if they completed therapy for the malignancy, are disease free from the malignancy for > 5 years, and are considered by their physician to be at < 30% risk of relapse
* No significant history of uncontrolled cardiac disease including, but not limited to, any of the following:

  * Uncontrolled hypertension
  * Unstable angina
  * Recent myocardial infarction (within the past 6 months)
  * Uncontrolled congestive heart failure
* No active bacterial, fungal, or viral infection
* No known HIV infection or active hepatitis B and/or hepatitis C infection
* No other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the study results

PRIOR CONCURRENT THERAPY:

* No concurrent biologic therapy, chemotherapy, or other antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12-12 (Actual); Primary Completion 2011-07-29 (Actual); Study Completion 2011-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig C. Hofmeister, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevnar: The conjugate vaccine for Streptococcus pneumoniae will be administered during weeks 9, 17, and 25 after autologous HSCT - the study nurse will arrange for the vaccine to be administered at the specified time and the patient will be instructed to notify an investigator or study nurse of any side effects of vaccine administration. At the specified times, patients will fill out the quality-of-life assessment. All patients enrolled on this trial will have samples procured for all proposed laboratory correlative studies.
  Streptococcus pneumoniae: Patients will receive 0.5 mL Prevnar in the deltoid muscle during weeks 9, 17, and 25 after autologous hematopoietic stem cell transplantation (HSCT)
  laboratory correlative studies: Approximately 30-mL of blood will be collected and sent to the appropriate research lab(s) for processing.
  quality-of-life assessment: Responses to Hospital Anxiety and Depression Scale, 9-item brief fatigue inventory 57, brief pain inventory, and the FACT-G.
Period: Overall Study
Arm/Group | Prevnar
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prevnar
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 51 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Immune Reconstitution
Description: Immune reconstitution as measured by response to conjugate vaccine to Streptococcus pneumoniae (Prevnar, PCV7), NK cell activity against autologous lymphoblastoid cell lines, and CMV & EBV tetramer responses after autologous transplant for myeloma
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Prevnar
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Serial Assessment of the Absolute Number of Circulating Regulatory T-cells and the Function of These Cells as Measured by Their Expression of TGFβ and Interleukin-10 (IL-10)
Time Frame: Up to 3 years
Population: Inadequate material collected to perform these assays
Arm/Group | Prevnar
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of Quality of Life With Inflammatory Cytokine Production of Peripheral Blood Monocytes
Time Frame: Up to 3 years
Population: Quality of Life surveys were not completed
Arm/Group | Prevnar
Number analyzed (Participants) | 0

4. Secondary Outcome: Quality of Life, Including Brief Pain Inventory
Description: The Brief Pain Inventory - Short Form (BPI-SF) asks respondents to rate the severity of their current, least, average, and worst pain over the previous 24 hours on a scale of 0 to 10. The BPI-SF also asks respondents to rate on a scale of 0 to 10 the degree to which pain interfered with seven different areas of their life (e.g., general activity, normal work, etc.)Scale 0-10 with 0 being no pain and 10 being pain as bad as you can imagine.
Time Frame: Up to 3 years
Population: Not all patients data was available due to incomplete surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevnar
Number analyzed (Participants) | 13
units on a scale | 2.8 (2.1)

5. Secondary Outcome: Quality of Life, Including Fatigue
Description: Brief Fatigue Inventory is a 9-item BFI assessing the severity of fatigue and the impact of fatigue on daily function. Scale 0-10 with 0 being no fatigue and 10 being as bad as you can imagine.
Time Frame: Up to 3 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevnar
Number analyzed (Participants) | 30
units on a scale | 2.55 (2.21)

6. Secondary Outcome: Collection of Baseline Immune Reconstitution and Quality of Life Pilot Data for Comparison in Future Post-transplant Immunotherapy Trials
Time Frame: Up to 3 years
Population: Data was not collect and analyzed for reporting purposes
Arm/Group | Prevnar
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Prevnar: The conjugate vaccine for Streptococcus pneumoniae will be administered during weeks 9, 17, and 25 after autologous HSCT - the study nurse will arrange for the vaccine to be administered at the specified time and the patient will be instructed to notify an investigator or study nurse of any side effects of vaccine administration. Streptococcus pneumoniae: Patients will receive 0.5 mL Prevnar in the deltoid muscle during weeks 9, 17, and 25 after autologous hematopoietic stem cell transplantation (HSCT)
Arm/Group | Prevnar
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevnar (N=30)
Infection with unknown ANC (Infections and infestations) | 23 (23) — Upper Respiratory Infection
Infection with unknown ANC (Infections and infestations) | 3 (3) — Pneumo fever with origin unknown
Fever with unknown origin (General disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes